CLINICAL TRIAL: NCT00401466
Title: Remote Follow-up for ICD-Therapy in Patients Meeting MADIT II Criteria (REFORM)
Brief Title: Remote Follow-up of Patients Receiving Implantable Cardioverter Defibrillator for Prophylactic Therapy
Acronym: REFORM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Jochen Proff, Biotronik SE & Co. KG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS024
Record Dates: First submitted 2006-11-17; First posted 2006-11-20 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2008-07

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia
Keywords: prophylactic ICD therapy; home monitoring; follow-up interval; remote follow-up
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Prolonged follow-up intervals every 12 months
  Interventions: Device: Implantable Cardioverter Defibrillator
- 2 (Active Comparator): Standard follow-up intervals of 3 months
  Interventions: Device: Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator — ICD with Biotronik Home Monitoring capability
  Other Names: Lexos VR-T, Lexos DR-T, Belos DR-T, Lumos VR-T

SUMMARY:
The completed MADIT II study has shown that implantation of a cardioverter-defibrillator (ICD) in patients with a reduced left ventricular ejection fraction and a prior myocardial infarction reduces death from any cause. The probability of the first therapy due to ventricular tachyarrhythmia was about 34% within 3 years. With a 3-month ICD-follow-up scheme, as it is in the standard ICD therapy, the majority of patients is followed more closely than necessary with respect to anti-tachyarrhythmia ICD therapy.

A Home Monitoring (HM) function has been integrated into several ICD models from Biotronik (Berlin , Germany), for close remote monitoring of ICD patients. The HM function may substitute in-clinic follow-up controls.

The objective of our study is to compare a standard 3-month follow-up scheme and a 12-month follow-up scheme using HM in ICD recipients with the "MADIT II indications". The comparison should be made with respect to the difference in follow-up burden and the associated costs, and regarding possible impact of the remote follow-up via HM on all cause mortality, hospitalization, and patients' quality of life.

DETAILED DESCRIPTION:
The completed MADIT II study has shown that implantation of a cardioverter-defibrillator (ICD) in patients with a reduced left ventricular ejection fraction and a prior myocardial infarction reduces death from any cause. The probability of the 1st therapy due to ventricular tachyarrhythmia was about 34% within 3 years, with an increasing incidence from year 1 to 3. With a 3-month ICD-follow-up scheme, as it is in the standard ICD therapy, the majority of patients is followed more closely than necessary with respect to anti-tachyarrhythmia ICD therapy.

A Home Monitoring (HM) function has been integrated into several ICD models from Biotronik (Berlin , Germany), for close remote monitoring of ICD patients. The HM function automatically transmits predefined parameters on a daily basis from the implanted devices to a web-based platform accessible only by registered patients' physicians. These data may substitute in-clinical follow-up controls.

The objective of our study is to compare a standard 3-month follow-up scheme and a 12-month follow-up scheme using HM in ICD recipients with the "MADIT II indications". The comparison should be made with respect to the difference in follow-up burden and the associated costs, and regarding possible impact of the remote follow-up via HM on all cause mortality, hospitalization, and patients' quality of life.

The patients should receive single- or dual-chamber ICD models with the HM function.

The pre-hospital-discharge protocol comprises standard ICD follow-up + specific ICD programming, and activation of the HM function. The 1st standard follow-up visit is performed 3 months after the pre-discharge control. At this visit the patients are randomized to 3- vs. 12-month follow-up scheme. For the 3-month follow-up group, routine visits are scheduled at 6, 9, 12, 15, 18, 21, 24, and 27 months after patient discharge. For the 12-month (remote) follow-up group, routine visits are scheduled at 15 and 27 months after discharge. In either group, additional visits are scheduled on patient demand, due to device or lead problems, or due to the following Cardio Report (Home Monitoring) findings: Elective ICD replacement point, the 1st shock after discharge, an ineffective shock, ineffective anti-tachycardia pacing, ventricular pacing impedance outside the pre-defined range, shock impedance lower than 25 Ohm or greater than 110 Ohm, frequent arrhythmia episodes (according to pre-specified criteria).

ELIGIBILITY:
Inclusion Criteria:

Indication for implantation of an implantable cardioverter-defibrillator (ICD) according to the patient selection criteria used in the MADIT-II trial:

* Myocardial infarction 1 month or more prior to entry
* Ejection fraction of 30% or less within 3 months before entry

Exclusion Criteria:

* NYHA functional class IV
* Coronary revascularization later than 5 days after ICD implantation
* First myocardial infarction within the past month
* Advanced cerebrovascular disease
* Any condition with a likelihood of death within the next 12 months
* Pacing indication
* Conventional ICD indication (i.e., criteria other than MADIT II)
* Living in an area with insufficient GSM coverage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Number of follow-up visits | 27 months

SECONDARY OUTCOMES:
Total costs | 27 months
Mortality from any cause | 27 months
Quality of life (SF-36) | 27 months
Hospitalization | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof. Dr., Study Chair — Herzzentrum Leipzig, Germany
Locations (5):
- Czechia (2):
  - Institute of clinical and experimental medicine, Prague
  - Hospital Na Homolce, Prague
- Germany (3):
  - Zentralklinik Bad Berka, Bad Berka
  - Herz- und Gefäßklinikum Bad Neustadt GmbH, Bad Neustadt an der Saale
  - Herzzentrum der Universität Leipzig, Leipzig

REFERENCES:
- [Result] Elsner C, Sommer P, Piorkowski C, Taborsky M, Neuser H, Bytesnik J, Geller J, Kottkamp H, Wiesmeth H, Hindricks G. A prospective multicenter comparison trial of Home Monitoring against regular follow-up in MADIT II patients: additional visits and cost impact. Comput Cardiol 33: 241-244, 2006.
- [Derived] Hindricks G, Elsner C, Piorkowski C, Taborsky M, Geller JC, Schumacher B, Bytesnik J, Kottkamp H. Quarterly vs. yearly clinical follow-up of remotely monitored recipients of prophylactic implantable cardioverter-defibrillators: results of the REFORM trial. Eur Heart J. 2014 Jan;35(2):98-105. doi: 10.1093/eurheartj/eht207. Epub 2013 Jul 18. PMID 23868932